CLINICAL TRIAL: NCT02178878
Title: Genetic and Demographic Factors That Influence the Pain and Progress of Labor
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: 17054
Record Dates: First submitted 2014-04-30; First posted 2014-07-01 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Rapid Progress of Labor
Keywords: Labor pain and progress, variation, genetic
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample for DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Progress, Pain: Progress, Pain
  Interventions: Genetic: Progress, Pain

INTERVENTIONS:
Genetic: Progress, Pain — Progress, Pain

SUMMARY:
The purpose of this study is to try to understand why the experience of labor differs among women. The investigators want to understand why some women have longer or shorter labors and why the amount of pain women experience is different. The investigators hope to be able to consider women more individually in terms of their pain and progress of labor.

DETAILED DESCRIPTION:
There is enormous variability among women in the progress of normal labor. Labor requires complex integrated interplay between the decidua, uterine cervix and myometrium that can take minutes, days or weeks to occur and is incompletely understood. Understanding the biological variables that underlie differences in labor progress has been hampered by the lack of appropriate models that allow sensitive statistical analysis. Identification of genetic and physiognomic factors that impact normal labor progress will allow for individualization of labor management and better use of societal resources.

Structural models of labor progress were first proposed by Friedman in the 1950s at Columbia University. Aspects of Friedman's model, such as the deceleration phase, have been debated since that time but Friedman's model allowed for identification and quantification of the latent and active phase of labor in populations. These concepts have been modified by the World Health Organization as the WHO Partogram, the use of which has resulted in reduced requirement of oxytocin and reduced incidence of cesarean section.

Dr. Flood's group has developed a continuous bi-exponential model of labor progress and sigmoidal model for labor pain that the investigators have statistically and experimentally validated in several independent databases. The investigators model can be used both prospectively in an individual labor and with large cohorts to identify variables that significantly affect the progress of labor.

The investigators have found in a previous work that parturients who carry G at the 27th amino acid beta-2 adrenergic receptors (β2AR) developed labor pain more rapidly that parturients with the common allele [1]. and the investigators also have found that catechol-O-methyltransferase (COMT) rs4633 genotype TT resulted in a slower latent phase rate, and oxytocin receptor rs53576 genotype GG transitioned to active labor earlier [2].

In this new project, the investigators are planning to use bigger data base, to detect further genes associations, and tested some pharmacogenetic variations that could explain the different response to same medications and doses among patients.

ELIGIBILITY:
Inclusion Criteria:

* Study participants will be women presenting in term labor.
* Patients of all ethnicities will be included.
* All subjects will be greater than or equal to 18 years of age and able to give consent.

Exclusion Criteria:

* Include preexisting pain syndromes or the regular taking of pain medications.
* Preterm birth (< 37 weeks) and preeclampsia.
* Cervical dilatation more than 6 cm

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant in active labor
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Labor progress variability | We will monitor data from the entire period of labor, which may last from 1-30 hours

SECONDARY OUTCOMES:
Respond variability to different induction, augmentation and pain management medication Prostaglandine, Oxytocin, Epidural analgesia | admission to hospital discharge ( est. 2-3 days)

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah S Terkawi, M.D., Principal Investigator — University of Virginia; Marcel E Durieux, M.D., Ph.D, Principal Investigator — University of Virginia; Pamela D Flood, M.D., Ph.D, Principal Investigator — Stanford University
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Terkawi AS, Jackson WM, Thiet MP, Hansoti S, Tabassum R, Flood P. Oxytocin and catechol-O-methyltransferase receptor genotype predict the length of the first stage of labor. Am J Obstet Gynecol. 2012 Sep;207(3):184.e1-8. doi: 10.1016/j.ajog.2012.06.079. Epub 2012 Jul 10. PMID 22939719
- [Background] Terkawi AS, Jackson WM, Hansoti S, Tabassum R, Flood P. Polymorphism in the ADRB2 gene explains a small portion of intersubject variability in pain relative to cervical dilation in the first stage of labor. Anesthesiology. 2014 Jul;121(1):140-8. doi: 10.1097/ALN.0000000000000258. PMID 24714117